CLINICAL TRIAL: NCT00837317
Title: Comparative Effect Of Different Oils For Frying On The Endothelial Function, The Oxidative Stress And The Postprandial Inflammatory Response
Brief Title: Different Oils For Frying and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Francisco Perez Jimenez, Reina Sofia University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Oils&Frying
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Endothelial Dysfunction
Keywords: Phenols; Laser-Doppler; Olive Oil; Sunflower Oil; Dimethylpolysiloxane; Postprandial; Inflammation; Oxidative Stress
MeSH Terms: conditions — Inflammation | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All the volunteer subjects will be administered four breakfast meals that have been prepared with four different types of oil, each of which will have been subjected to a standardised frying. The meals will be administered according to a cross-randomized Latin squares design
  Interventions: Dietary Supplement: Olive Oil, SF, SF+DMP, SF+phenols

INTERVENTIONS:
Dietary Supplement: Olive Oil, SF, SF+DMP, SF+phenols — All the volunteer subjects will be administered four breakfast meals that have been prepared with four different types of oil, each of which will have been subjected to a standardised frying. The meals will be administered according to a cross-randomized Latin squares design
  Other Names: SF=Sunflower Oil; DMP=dimethylpolysiloxane

SUMMARY:
The purpose of this study is to compare the effects of the consumption of different oils (olive oil, sunflower oil, sunflower plus dimethyl-polysiloxane, sunflower plus phenols) previously submitted to heating in postprandial endothelial function, inflammation and oxidative stress in healthy young men.

DETAILED DESCRIPTION:
To determine whether the consumption by healthy persons of an oil exposed to high temperatures, designed to have a composition of healthy fats (predominantly monounsaturated fats and with less than 10% palmitic acid) and to contain an abundance of antioxidants typically found in olive oil (phenolic compounds), will improve the vasodilatory response that depends on the endothelium, and buffer the inflammatory and postprandial oxidative response that is produced by the oils that are being used ever more frequently for frying purposes (sunflower oil and oil to which butylated hydroxytoluene (BHT) has been added), using virgin olive oil exposed to the same heating regime as a reference oil.

ELIGIBILITY:
Inclusion Criteria:

* Investigators will select obese people (BMI ranged 25 to 40).

Exclusion Criteria:

* Evidence of malignancy or severally ill (life expectancy lesser than 5 years).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent postprandial vasodilatation measured by laser-doppler after the consumption of 4 different oils: -Virgin Olive Oil -Sunflower Oil -Sunflower High Oleic plus phenols -Sunflower High Oleic plus dimethylpolysiloxane | 0, 2, 4 hours after the meals

SECONDARY OUTCOMES:
Assessment of pro-oxidative state, as evaluated via the determination of F2 isoprostane, nitrates and nitrites, total plasma antioxidative capacity, lipoperoxides and oxidised proteins. | 0 and 4 hours after the meal
Assessment of proinflammatory state in both soluble plasma markers (IL-6, TNF-alpha, MCP-1, VCAM-1, ICAM-1) and the postprandial activation (RNAm) of IL-6, TNF-alpha, Rel-A, I-kappaB-alpha, MIF, MMP-9 y MCP-1 genes. | 0 and 4 hours after the meal
Assessment of interrelationship of postprandial lipaemic response and the response of the inflammatory markers and of the oxidative metabolism with each of the oils employed in the study. | 0, 4 hours after the meal

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Perez-Jimenez, MD, PhD, Principal Investigator — Reina Sofia University Hospital
Locations (1):
- Reina Sofia University Hospital, Córdoba, Cordoba, Spain

REFERENCES:
- [Derived] Perez-Herrera A, Delgado-Lista J, Torres-Sanchez LA, Rangel-Zuniga OA, Camargo A, Moreno-Navarrete JM, Garcia-Olid B, Quintana-Navarro GM, Alcala-Diaz JF, Munoz-Lopez C, Lopez-Segura F, Fernandez-Real JM, Luque de Castro MD, Lopez-Miranda J, Perez-Jimenez F. The postprandial inflammatory response after ingestion of heated oils in obese persons is reduced by the presence of phenol compounds. Mol Nutr Food Res. 2012 Mar;56(3):510-4. doi: 10.1002/mnfr.201100533. Epub 2011 Dec 9. PMID 22162245